CLINICAL TRIAL: NCT01390701
Title: Blood Pressure Lowering Effect of Low-frequency Transcutaneous Electrical Nerve Stimulation and Felodipin
Brief Title: Blood Pressure Lowering Effect of Transcutaneous Electrical Nerve Stimulation
Acronym: HyperTENSion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Jonas Silverdal MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HyperTENSion
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: randomized; cross-over; transcutaneous electrical nerve stimulation; felodipin; hypertension; blood pressure; treatment
MeSH Terms: conditions — Hypertension | interventions — Transcutaneous Electric Nerve Stimulation; Felodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcutaneous electr. nerve stimulation (Experimental)
  Interventions: Device: transcutaneous electrical nerve stimulation
- felodipin (Active Comparator)
  Interventions: Drug: felodipin

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation — 30 min of bi-daily low-frequency transcutaneous electrical nerve stimulation on the upper extremities. Duration: 28+-4 days.
  Other Names: 2 Hz Primo Pro stimulators (CefarCompex, Sweden).
  Arms: transcutaneous electr. nerve stimulation
Drug: felodipin — 2,5mg of felodipin once daily. Duration: 28+-4 days.
  Arms: felodipin

SUMMARY:
The purpose of this study is to compare the blood pressure reducing property of transcutaneous electrical nerve stimulation with the blood pressure reducing drug felodipin.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for development of several vascular complications and is common world wide. Drug treatment is often necessary to achieve adequate blood pressure reduction but blood pressure control in studied countries is unsatisfactory low. Reasons for failure in treatment are several. Among others reasons intolerable side-effects may prevent successful treatment irrespective of the number of drugs.

Transcutaneous electrical nerve stimulation (TENS) constitutes no risk of interaction with pharmacological agents and previous studies have reported blood pressure reduction.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hypertension, untreated or currently treated with a maximum of one blood pressure (BP) lowering agent

Exclusion Criteria:

* systolic blood pressure >170 mmHg and/or diastolic blood pressure of >105 mmHg
* second- or third-degree atrioventricular block
* current use of opiates or other intoxicants
* neurological disorders (such as Parkinson's disease, multiple sclerosis or peripheral neuropathy)
* need of treatment with TENS, regardless the reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | four weeks
  Office blood pressure measurement and 24-h ambulatory blood pressure monitoring after four week periods of treatment in a cross-over design with intervening four week washout and subsequent four week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Silverdal, MD, Principal Investigator — Department of Medicine, Geriatrics and Emergency Medicine, Sahlgrenska University Hospital/Östra; Karin Manhem, ass.prof., Principal Investigator — Institute of Medicine, Department of Emergency and Cardiovascular Medicine, Sahlgrenska University Hospital/Sahlgrenska; Clas Mannheimer, professor, Principal Investigator — Multidisciplinary Pain Center, Sahlgrenska University Hospital/Östra; Georgios Mourtzinis, MD, Principal Investigator — Department of Medicine, Sahlgrenska University Hospital/Mölndal; Elisabet Stener-Victorin, ass.prof., Principal Investigator — Institute of Neuroscience and Physiology, Department of Physiology, University of Gothenburg
Locations (1):
- Department of Medicine, Geriatrics and Emergency Medicine, Sahlgrenska University Hospital/Östra, Gothenburg, Sweden